CLINICAL TRIAL: NCT07285915
Title: Stress as a Key Factor Influencing the Onset and Course of Cardiac Arrest
Brief Title: The Role of Stress in Cardiac Arrest (Cortizol CPR)
Acronym: Cortizol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Pilsen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Stress
Record Dates: First submitted 2025-11-18; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Chronic Stress; Cardiac Arrest (CA); Post-Resuscitation Syndrome; Heart Attack
Keywords: cardiac arrest; chronic stress; kortizol; hair
MeSH Terms: conditions — Heart Arrest; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac arrest (Experimental): Cardiac arrest
  Interventions: Diagnostic Test: Sample of hair
- Heart attack (Experimental): Heart attack
  Interventions: Diagnostic Test: Sample of hair

INTERVENTIONS:
Diagnostic Test: Sample of hair — Sampling of 3cm of hair due to level of cortizol.

SUMMARY:
The aim of this study is to assess long-term stress in patients after an out-of-hospital cardiac arrest. To do this, we will measure levels of the stress hormone cortisol in hair samples. Cortisol is produced in larger amounts during periods of ongoing stress and builds up in the hair as it grows. Because hair grows about 1 cm per month, a 3 cm hair sample can show your average stress level over the past three months. The results will be compared with anonymized information from your medical records and the care you received before and during your hospital stay.

DETAILED DESCRIPTION:
Despite significant advances in resuscitation medicine, out-of-hospital cardiac arrest (OHCA) continues to carry a poor prognosis, with survival accompanied by good neurological outcomes in only about 30% of cases. In Europe, OHCA affects approximately 67-170 individuals per 100,000 annually; in the Czech Republic, the incidence is around 90 per 100,000. Most cardiac arrests (60-70%) are of cardiovascular origin, where long-term stress is a known contributing risk factor.

Chronic stress not only influences the development of cardiovascular disease but also affects its clinical manifestation by modulating the autonomic nervous system-an essential regulator of heart rhythm and arrhythmogenic risk. Therefore, it is plausible that prolonged stress also contributes to the onset and course of cardiac arrest.

While the relationship between chronic stress and cardiovascular disease has been well documented, data specifically linking stress to out-of-hospital cardiac arrest are still lacking. The pathophysiological factors influencing the onset and refractoriness of OHCA also remain unclear.

This study aims to evaluate chronic stress levels in patients after OHCA by measuring cortisol concentrations in hair samples. Since cortisol accumulates in hair during its growth, a 3 cm segment reflects stress exposure over the previous three months. These findings will be correlated with patients' demographic and clinical profiles, including post-resuscitation condition severity, neurological outcomes, and potential arrest refractoriness.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest
* Heart attack
* 18 - 100 years

Exclusion Criteria:

* Disapproval patient´s relatives with the study
* Chronical treatment with corticoids and antidepresives

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Hair cortisol levels assessment in CA patients vs heart attack patients | Enrollment
  Hair cortisol levels assessment in CA patients vs heart attack patients

SECONDARY OUTCOMES:
Correlation of neurological outcomes using the CPC scale in CA patients with hair cortisol levels. | 30 and 90 days after CA
  Correlation of neurological outcomes using the CPC scale in CA patients with hair cortisol levels.
Correlation between the severity of the post-resuscitation course according to the severity of organ damage (heart, lung, kidneys, brain ) and hair cortisol levels | 30 days after CA
  Correlation between the severity of the post-resuscitation course according to the severity of organ damage (heart, lung, kidneys, brain ) and hair cortisol levels

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Pilsen, Pilsen, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No